CLINICAL TRIAL: NCT01580657
Title: Experimental Analysis of HIV Risk Assessment Reactivity in South African Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: PRO00005529; 5R01MH077515-04 (NIH)
Record Dates: First submitted 2012-04-12; First posted 2012-04-19 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2012-04

CONDITIONS: HIV Prevention and Assessment Reactivity
Keywords: HIV; Prevention; Methods; Assessment reactivity; South Africa; Youth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Detailed baseline interview, enhanced HIV intervention (Experimental): Participants in this group will receive a detailed sexual behavior interview, similar to measures used in major intervention trials. This measure will identify the instances in which participants engaged in sexual behaviors with specific partners during a 90 day retrospective reporting period. Participants will then complete an empirically validated 60-minute session HIV-risk reduction intervention (Simbayi, Kalichman, Skinner et al., 2004) consisting of exercises to increase HIV/AIDS knowledge, motivation to reduce risk, behavior self-management skills, and sexual communication skills and reduce HIV-related stigma.
  Interventions: Behavioral: Detailed baseline interview, enhanced HIV intervention
- General baseline interview, enhanced HIV intervention (Experimental): Participants in this group will receive the same procedures as in (A) except that the behavioral measure will consist of single-item frequency questions regarding sexual behaviors during the prior 90 days, questions that do not lead the participant to focus on specific instances of behavior.
  Interventions: Behavioral: General baseline interview, enhanced HIV intervention
- No baseline interview, enhanced HIV intervention (Experimental): This group will receive the same enhanced intervention procedures as in (A) and (B), but they will not be interviewed at baseline.
  Interventions: Behavioral: No baseline interview, enhanced HIV intervention
- D. Detailed baseline interview, standard of care intervention (Active Comparator): Participants in this group will receive the same interview procedure as in (A) but instead of the enhanced intervention, They will undergo the standard clinical exam and health education that at the Spencer Rd. Clinic.
  Interventions: Behavioral: Detailed baseline interview, standard of care intervention
- E. General baseline interview, standard of care intervention (Active Comparator): Participants in this group will complete the general baseline interview described in (B) and then receive the standard care at the clinic.
  Interventions: Behavioral: General baseline interview, standard of care intervention
- F. No baseline interview, standard of care intervention (Active Comparator): Participants assigned to this group will be consented on the day they are recruited, but will not receive further study contact on that day other than being scheduled to return for follow up assessments.
  Interventions: Behavioral: No baseline interview, standard of care intervention

INTERVENTIONS:
Behavioral: Detailed baseline interview, enhanced HIV intervention — Participants in this group will receive a detailed sexual behavior interview, similar to measures used in major intervention trials. This measure will identify the instances in which participants engaged in sexual behaviors with specific partners during a 90 day retrospective reporting period. Participants will then complete an empirically validated 60-minute session HIV-risk reduction intervention (Simbayi, Kalichman, Skinner et al., 2004) consisting of exercises to increase HIV/AIDS knowledge, motivation to reduce risk, behavior self-management skills, and sexual communication skills and reduce HIV-related stigma.
  Arms: Detailed baseline interview, enhanced HIV intervention
Behavioral: General baseline interview, enhanced HIV intervention — Participants in this group will receive the same procedures as in (A) except that the behavioral measure will consist of single-item frequency questions regarding sexual behaviors during the prior 90 days, questions that do not lead the participant to focus on specific instances of behavior.
  Arms: General baseline interview, enhanced HIV intervention
Behavioral: No baseline interview, enhanced HIV intervention — This group will receive the same enhanced intervention procedures as in (A) and (B), but they will not be interviewed at baseline.
  Arms: No baseline interview, enhanced HIV intervention
Behavioral: Detailed baseline interview, standard of care intervention — Participants in this group will receive the same interview procedure as in (A) but instead of the enhanced intervention, They will undergo the standard clinical exam and health education that at the Spencer Rd. Clinic.
  Arms: D. Detailed baseline interview, standard of care intervention
Behavioral: General baseline interview, standard of care intervention — Participants in this group will complete the general baseline interview described in (B) and then receive the standard care at the clinic.
  Arms: E. General baseline interview, standard of care intervention
Behavioral: No baseline interview, standard of care intervention — Participants assigned to this group will be consented on the day they are recruited, but will not receive further study contact on that day other than being scheduled to return for follow up assessments.
  Arms: F. No baseline interview, standard of care intervention

SUMMARY:
Randomized clinical trials of HIV prevention interventions typically include extensive baseline assessments of the risk behaviors that interventions target. Such pretests have the potential to direct participants' attention to the factors that put them at risk of HIV infection. Evidence from intervention study control groups, the motivational enhancement and attitude change literature, and our preliminary studies suggest that assessments that lead people to think about behaviors with potentially negative outcomes lead to motivation for risk behavior reduction. As a consequence, HIV intervention research using baseline assessments may not accurately predict the impact of a given HIV prevention intervention outside of the research context, in particular when interventions are evaluated among high-risk, isolated individuals. However, the actual effects as well as public-health consequences and mechanisms of HIV assessment reactivity have never been systematically tested.

The proposed assessment reactivity study will be conducted in South Africa, a country with high levels of HIV prevalence, incidence, and stigma. The Republic of South Africa's HIV/AIDS epidemic has emerged recently relative to other sub-Saharan countries, and yet 21.5% of South Africans aged 15-49 -- more than 1 in 5 people -- are infected with HIV (UNAIDS, 2004). Despite the common presence of HIV in South Africa, it remains largely a hidden disease and HIV-related stigma interferes with peoples' ability to protect themselves through open discussion or spontaneous reflection on personal risk. Under these conditions, it is reasonable to expect a sizable effect from directing people's attention to their HIV relevant behaviors, an effect that could be incorrectly ascribed to brief interventions used in low-resource settings. The conditions in South Africa, therefore, heighten the clinical and public health significance of the assessment reactivity issue in that (a) it is vital to understand how reactivity may affect the results of behavioral intervention trials, and (b) it may be possible to capitalize on assessment reactivity through brief, assessment-based interventions.

This study will allow us to achieve our primary aim:

1. To separate the effect of a brief HIV-risk reduction intervention from the potential effects of two types of baseline assessment commonly applied in HIV intervention research: a detailed, calendar-based assessment and a general frequency assessment. The detailed calendar-based assessment will potentially lead participants to observe themselves in specific risk-behavior situations, providing them with the opportunity to reassess the risk involved in those situations in light of their health goals and thus motivating them for behavior change. The general frequency assessment will merely prompt participants to estimate the overall frequency with which they engaged in several HIV-related behaviors. The effect of these assessments on participants' sexual behavior will be examined alone and in combination with the HIV-risk reduction intervention.

In addition, this project has two important secondary aims:

1. To generate urgently needed additional efficacy data for a promising HIV risk reduction intervention culturally tailored for use and found to be effective in South Africa
2. To determine potential HIV preventive effects of different types of HIV risk behavior assessments on risk behavior reduction in South Africa for future intervention development

To achieve the above aims, the investigators will:

1. Recruit 1500 patients (50% women), age 18-44, from the Spencer Rd. STD Clinic, Cape Town, South Africa.
2. Randomly assign participants within gender to one of 6 study arms in a modified Solomon Four-Group (SFG) design. The 2 (intervention: standard of care vs. an efficacious theory based HIV prevention intervention) x 3 (baseline face-to-face interview: none vs. basic single-item frequency questions vs. detailed partner-by-partner calendar-based interview) factorial design is depicted below:

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* presenting at the site B youth STD clinic for STD services, and
* residence within the clinic's catchment area.

Exclusion Criteria:

* The exclusion criteria will be a previous HIV-positive diagnosis or
* Testing HIV-positive on the day of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1728 (Actual)
Dates: Start 2006-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Reactivity assessment | Three month follow up
  Using the analytic strategy for the SFG design, we will use the follow-up data point to test our hypotheses that there will be a significant interaction between assessment conditions x intervention conditions.
  Analyses will explore the effects of assessment and intervention on the factors presumed to mediate the effect of assessment reactivity (increases in perceived risk and safer sex intentions). Moderator analyses will observe if type of assessment interacts with the level of reported risk behavior (dichotomized as low and high).

SECONDARY OUTCOMES:
Risk Behavior Frequency | Baseline and three month follow up
  1. To separate the effect of a brief HIV-risk reduction intervention from the potential effects of two types of baseline assessment commonly applied in HIV intervention research: a detailed, calendar-based assessment and a general frequency assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lance S Weinhardt, PhD, Principal Investigator — Medical College of Wisconsin and UW Milwaukee Zilber School of Public Health
Locations (1):
- Site B Youth Clinic, Khayelitsha, South Africa

REFERENCES:
- [Background] Kalichman SC, Cain D, Weinhardt L, Benotsch E, Presser K, Zweben A, Bjodstrup B, Swain GR. Experimental components analysis of brief theory-based HIV/AIDS risk-reduction counseling for sexually transmitted infection patients. Health Psychol. 2005 Mar;24(2):198-208. doi: 10.1037/0278-6133.24.2.198. PMID 15755234
- [Background] Kalichman SC, Rompa D, Coley B. Experimental component analysis of a behavioral HIV-AIDS prevention intervention for inner-city women. J Consult Clin Psychol. 1996 Aug;64(4):687-93. doi: 10.1037//0022-006x.64.4.687. PMID 8803358
- [Background] Weinhardt LS, Carey KB, Carey MP. HIV risk sensitization following a detailed sexual behavior interview: a preliminary investigation. J Behav Med. 2000 Aug;23(4):393-8. doi: 10.1023/a:1005505018784. PMID 10984867
- [Background] Weinhardt LS. Effects of a detailed sexual behavior interview on perceived risk of HIV infection: preliminary experimental analysis in a high risk sample. J Behav Med. 2002 Apr;25(2):195-203. doi: 10.1023/a:1014888905882. PMID 11977438
- [Background] Weinhardt LS, Forsyth AD, Carey MP, Jaworski BC, Durant LE. Reliability and validity of self-report measures of HIV-related sexual behavior: progress since 1990 and recommendations for research and practice. Arch Sex Behav. 1998 Apr;27(2):155-80. doi: 10.1023/a:1018682530519. PMID 9562899